CLINICAL TRIAL: NCT02049710
Title: Randomized Controlled Trial Evaluating the Effectiveness of Interactive Video Interventions to Reduce Teen Pregnancy and Teen Automobile Injuries
Brief Title: Teen Video Study to Reduce Risky Driving and Sexual Behavior in Adolescents
Acronym: TVS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carnegie Mellon University (Other)
Collaborators: West Virginia University (Other); University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TPP-TVS-01; 5 TP1AH000040 (Other Grant/Funding Number: Office of Adolescent Health, HSS)
Record Dates: First submitted 2013-12-18; First posted 2014-01-30 (Estimated); Results first posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2021-06

CONDITIONS: Pregnancy; Sexually Transmitted Infections; Automobile Accidents
Keywords: pregnancy prevention, condom use, self efficacy
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sexual Behavior Intervention (Active Comparator): Video based intervention based on changing risky behavior associated with sexual behavior.
  Interventions: Behavioral: Seventeen Days
- Driving behavior intervention (Active Comparator): Video based intervention based on changing risky behavior associate with driving
  Interventions: Behavioral: Driving Skills for Life

INTERVENTIONS:
Behavioral: Seventeen Days — Interactive video includes highlighting salience of active choices in sexual decision making, modeling different responses to sexual situations, cognitive rehearsal of preventive behaviors, and information about hormonal and non-hormonal contraception
  Arms: Sexual Behavior Intervention
Behavioral: Driving Skills for Life — Interactive video includes guidance and practice for safe driving techniques, driver and car care tips, an eco-driving learning module, and interactive driving games.
  Arms: Driving behavior intervention

SUMMARY:
The purpose of this study is to measure the effects of an interactive video on adolescent risky behaviors and outcomes, with one video intended to reduce teen pregnancies and the other intended to reduce automobile accidents.

DETAILED DESCRIPTION:
Motor vehicle crashes cause one-third of teenage deaths and many serious injuries. Teen drivers ages 16 to 19 are four times more likely than older drivers to crash. Death and injuries could be reduced with a change in behaviors that include improved visual and attention skills while driving, more seat belt use, appropriate speed control, and not combining drinking or texting with driving. Sexually transmitted infections (STIs) and unplanned pregnancies are particularly common among adolescents. The U.S. adolescent birthrate is by far the highest among industrialized nations. These problems can be decreased by less sexual activity and better protection.

This study uses a randomized controlled trial to measure how well interactive video interventions can reduce these common risks to adolescents. Adolescent females will be invited to participate if they are currently seeking care at a participating clinic. They will answer survey questions about their driving and sexual behaviors, and then a computer will determine whether they will be given a video about driving or a video about sexual behavior. Participants will have unlimited access to their video, which they can watch at their clinic or from any Internet-enabled computer, and will be followed for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient at participating healthcare facility
* Unmarried at time of enrollment
* Not pregnant at time of enrollment
* Available for contact over ensuing 6 months

Exclusion Criteria:

* Apparent or stated inability to comprehend consent or assent form (e.g., language barrier or cognitive ability)
* No ability to provide at least 2 methods of contact
* Married or pregnant at time of enrollment

Ages: 14 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Females only as the project is focusing on teen pregnancy prevention. (self-representation of gender)
Enrollment: 1317 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie S Downs, Ph.D., Principal Investigator — Carnegie Mellon University; Pamela J Murray, MD, MHP, Principal Investigator — West Virginia University
Locations (3):
- United States (3):
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - West Virginia University, Morgantown, West Virginia

REFERENCES:
- [Background] Downs JS, Ashcraft AM, Murray PJ, Berlan ED, Bruine de Bruin W, Eichner J, Fischhoff B, Leary JM, McCall RB, Miller E, Salaway J, Smith-Jones J, Sucato GS. Video Intervention to Increase Perceived Self-Efficacy for Condom Use in a Randomized Controlled Trial of Female Adolescents. J Pediatr Adolesc Gynecol. 2018 Jun;31(3):291-298.e2. doi: 10.1016/j.jpag.2017.10.008. Epub 2017 Nov 7. PMID 29126824

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized once they consented to participate and before the baseline survey.
Period: Overall Study
Arm/Group | Sexual Behavior Intervention | Driving Behavior Intervention
Started | 653 | 664
Completed | 334 | 340
Not Completed | 319 | 324
Not completed — Lost to Follow-up | 319 | 324

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sexual Behavior Intervention | Driving Behavior Intervention | Total
Number analyzed (Participants) | 653 | 664 | 1317
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 503 | 505 | 1008
  Between 18 and 65 years | 150 | 159 | 309
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 17.18 [14 to 19] | 17.25 [14 to 19] | 17.20 [14 to 19]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 653 | 664 | 1317
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 653 | 664 | 1317

OUTCOME MEASURES:

1. Primary Outcome: Perceived Self-efficacy for Condom Use
Description: To assess the effects of the Seventeen Days interactive video on young women's perceived self-efficacy for using condoms 6 months after being offered the intervention, relative to a control.
Time Frame: 6 months
Population: Sexually active female adolescents ages 14 to 19 years. The overall number of participants analyzed are those that completed the baseline survey, video component and the 6 month survey.
Measure: Mean (95% Confidence Interval); unit: summation score
Arm/Group | Sexual Behavior Intervention | Driving Behavior Intervention
Number analyzed (Participants) | 334 | 340
summation score | 13.00 [12.74 to 13.24] | 12.48 [12.15 to 12.74]
Statistical Analysis 1: Comparison: Sexual Behavior Intervention vs Driving Behavior Intervention; Summation scores are reported across 3 items measured on a 5-point scale from 1(not at all sure)to5(very sure), which loaded together on a principal components analysis of the baseline data.The summation score thus represents a theoretical range from 3 to 15.The 3 items were as follows:Indicate How Sure You are that You Would be Able to Perform Each of the Following:a)Get the money needed to buy condoms b)Walk into a store&buy condoms c)Find a place to get condoms for free(Cronbach alpha-0.72); Test type: Other; Mean Difference (Final Values) = 5.06, 95% CI 2-sided [3 to 15]

ADVERSE EVENTS:
Time Frame: 6 months per participant
Description: Low risk study - watching a video intervention on a computer/tablet.
Arm/Group | Sexual Behavior Intervention | Driving Behavior Intervention
All-Cause Mortality (participants affected / at risk) | 0/653 | 0/664
Serious Adverse Events (participants affected / at risk) | 0/653 | 0/664
Other Adverse Events (participants affected / at risk) | 0/653 | 0/664

LIMITATIONS AND CAVEATS:
Because this intervention was a pregnancy prevention strategy, we recruited participants at risk for pregnancy(ie, female adolescents with recent sexual activity)&presented content targeted at heterosexual sexual behavior. Therefore, these findings are, by design, not generalizable to adolescent women having sex only with other women or to male adolescents. High overall attrition rates before as well as after randomization might limit generalizability of the findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No